CLINICAL TRIAL: NCT02921958
Title: The Life Participation for Parents as an Outcome Measure
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0326
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2016-09

CONDITIONS: Parents
Keywords: Parents of children with disabilities
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: occupational therapy — Family-centered occupational therapy services

SUMMARY:
Data was collected from Parents of children who were receiving occupational therapy services. Three assessment tools were used: 1. Life Participation for Parents, 2. Infant Toddler Sensory Profile, and 3) Child Behavior Checklist. Data was used to pursue 2 investigations.

1. Is the Life Participation for Parents responsive to change after intervention?
2. Are there correlations between child behavior, child sensory processing, and parental participation in their own lives while raising a child with special needs.

DETAILED DESCRIPTION:
Introduction and Purpose:The Life Participation for Parents is an assessment tool designed to measure a parent's ability to participate in daily life while raising a child with special needs. Previous studies have established the effectiveness of the instrument in providing valuable information for designing family-centered goals and intervention. Further investigation is needed to determine if the instrument is sensitive enough to measure change after intervention. This study is designed to further develop the LPP as an assessment for providing family-centered intervention for children with special needs and their families and to investigate child characteristics leading to issues in parental participation.

Background: Parents raising children with special needs encounter many challenges in their daily lives. However, the initial studies using the LPP determined that these challenges cannot be predicted by age, gender, or diagnoses of the child, the time the child has been in therapy, or the age, gender, or marital status of the parent. These challenges are unique to each individual and therefore an instrument is needed to assess individual parental needs to facilitate family-centered intervention.Family-centered practice in pediatric occupational therapy involves working with parents, families, and the child with special needs to facilitate participation in life through engagement in occupation. Occupational therapy practitioners frequently interpret family-centered practice as parental involvement in establishing and facilitating child- related goals. However, family-centered practice goes beyond child-related goals to incorporate changing the quality of life for the whole family. Families are interdependent, and intervention with the child can have a significant impact on life participation for the entire family, especially the parents. Raising a child with special needs can influence a parent's time usage, health, and choice of activities. To provide best-practice family-centered intervention, therapists need to understand individual barriers to life participation for the child, parents, and other family members. The LPP is a 22 item self-report questionnaire using a 5 point Likert scale. Each item also has space for a qualitative comment regarding the response. It is designed to be used by clinical practitioners such as occupational therapists, physical therapists, or speech and language pathologists in determining issues parents are having in participating in their daily lives. The issues identified by the LPP can then initiate further conversations between parent and clinician and assist with developing family-centered intervention goals. The LPP was developed using an Occupational Adaptation frame of reference providing items on both the efficiency and the effectiveness of a parent's ability to participate in life activities effected by raising a child with special needs. A preliminary principle component analysis revealed evidence for the two subscales. The LPP takes approximately10 minutes to complete by the parent and is scored easily by the therapist. Two other questionnaires (Infant Toddler Sensory Profile and Child Behavior Checklist) will be used to further investigate the impact of child behaviors on parent participation. Occupational therapists treat numerous young children with sensory processing abnormalities due to developmental delays. Sensory processing is commonly understood to mean the process by which the brain receives and makes use of all forms (tactile, auditory, visual etc.) of sensations to generate behavioral responses to the environment. Research shows that between 45% and 96% of children with Autism Spectrum Disorders (ASDs) and other developmental disorders present with sensory abnormalities, and sensory-related behaviors often drive referrals to occupational therapy. The majority of research in this area focuses on school-age children with ASDs. The parents of these children identify increased levels of stress and disruption to family life and participation in routines as a result. Since family members are interdependent, each member's ability to participate in occupations affects their own health and the health of the others. There is virtually no research on how sensory abnormalities and sensory-driven behavior of young children (0-3 years-old) affect parent participation in occupations. This is a critical factor to occupational therapy intervention for young children and their families.3. Summary of Project:The proposed study will use a pretest - intervention - posttest longitudinal design to assess the sensitivity of the LPP to measure change. A previous study established that the responses on the LPP were static over the short term (2-3 weeks) when there was no focused intervention between pretest and posttest (Fingerhut, 2013). At pretest, parent participants with children under the age of 3 will also be asked to complete the Infant Toddler Sensory Profile (ITSP) and Child Behavior Checklist (CBCL). This information will be correlated with parent participation on the LPP to investigate the effect of these child characteristics on parent participation.4. Study Procedures:Occupational therapist participants will be recruited from pediatric occupational therapy clinics and early intervention programs throughout Texas. Occupational Therapists (OTs) (n=30) will be approached by the investigators to ask 2 parents from their current clients to complete the LPP (n=60). If these parents identify issues that the therapist believes would be amenable to family-centered intervention in a 3 month time frame the parents will be enrolled into the longitudinal study. If not the therapist will continue to recruit until they enroll 2 parents. Parents with children under the age of 3 will also be asked to complete the ITSP and CBCL at this initial stage. This information will be used to investigate the effect of measured child characteristics on parental participation. The parents with children under the age of 3 may also be enrolled into the longitudinal aspect of the study depending on the issues they describe on the LPP. Parents with children under the age of 3 will continue to be recruited until there are 50 participants.For parents recruited for the longitudinal aspect of the study, the therapist will use the information from the LPP to further explore the responses with the parents and then collaboratively establish one family-centered goal related to an item or items on the LPP. The therapist will then design intervention to address this goal in addition to the established intervention he or she was providing for the child and family. The study researchers will provide information on family-centered intervention, training, and strategies to assist the therapists in providing effective family-centered intervention.Intervention will be provided for three months or until the child's therapy is discontinued. At this point (3 months or discontinuation), the parent will complete the LPP again. The therapist will complete a short survey including the goal established, the intervention provided, and the observed outcome of the intervention. Therapists will also be interviewed regarding their experience using the LPP to facilitate family-centered intervention.

Data Analysis/ Study Questions1. Is there a significant positive change on the overall LPP score for those parent participants whose intervention outcome was described as positive by the therapist? (Wilcoxon signed ranks test). 2. Is there a significant positive change on the LPP Items most closely related to the established goals for those parent participants whose intervention outcome was described as positive by the therapist?(Wilcoxon signed ranks test).3. Do levels of sensory processing as measured by the Infant Toddler Sensory Profile (ITSP) correlate with parent participation as measured by LPP?4. Do levels of maladaptive behavior, as measured by the Child Behavior Checklist (CBCL) correlate to levels of parent participation as measured by the LPP?5. Does the pattern of sensory presentations as measured by the ITSP correlate with maladaptive behaviors as measured by CBCL?Study data (demographics and data) from LPP completion (pretest only for those in the longitudinal study) will be added to data from previous studies (n= 162 + 60plus) for confirmatory principle component analysis (oblique rotation).

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with disabilities receiving occupational therapy services who identify at least one family-centered goal that is amenable to OT intervention for the instrument responsiveness question.
* Parents of children under the age of 3 with sensory processing disabilities receiving occupational therapy services for the correlational questions

Exclusion Criteria:

* Do not meet above criteria

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children with disabilities receiving occupational therapy services.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Life Participation for Parents | 3 - 6 months intervention
  Pretest - post-test design to examine responsiveness properties of instrument

CONTACTS AND LOCATIONS:
Overall Officials: Pataricia E Fingerhut, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fingerhut PE. Life Participation for Parents: a tool for family-centered occupational therapy. Am J Occup Ther. 2013 Jan-Feb;67(1):37-44. doi: 10.5014/ajot.2013.005082. PMID 23245781
- [Background] Fingerhut PE. Measuring outcomes of family-centered intervention: development of the Life Participation for Parents (LPP). Phys Occup Ther Pediatr. 2009;29(2):113-28. doi: 10.1080/01942630902784795. PMID 19401926